CLINICAL TRIAL: NCT06629922
Title: Sensory Interaction and Balance Control During Standing and Walking Under Challenging Conditions in Healthy Young and Older Adults
Brief Title: Sensory Interaction and Balance Control During Standing and Walking in Healthy Young and Older Adults
Status: Not yet recruiting | Type: Observational
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Pieter Meyns, Assoc. Prof., Hasselt University
Other Study IDs: HasseltU100
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Healthy; Young Adults; Older Adults (65 Years and Older); Elderly
Keywords: sensory interaction; sensory reweighting; older adults; balance; fall risk; fall

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Young Adults: a) aged between 18 to 35 years old and, b) have never been diagnosed with somatosensory, visual, and vestibular deficits as reported by the participants
  Interventions: Other: No intervention
- Older Adults: a) are 65 years old and over and, b) have not fallen in the last 12 months will also be invited to participate
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a observational study and the participants will not receive any intervention

SUMMARY:
This project is designed to: a) develop a new test called UHasselt Locomotor Sensory Integration Test (UHLSINT) which would allow us to evaluate sensory interaction process in locomotion assess whether Locomotor CTSIB and to investigate whether UHLSINT is a reliable test to evaluate sensory interaction in both young and older adults, b) evaluate the difference in sensory interaction and balance performance between standing and walking between both young and older adults, c) examine the changes in sensory interaction process under challenging conditions such as perturbations, dual-task, and when both are present between both young and older adults, d) examine the association between overall fall risk defined by the single-large perturbations and sensory interaction processes used during all the trials in both age groups.

In order to achieve these aims, 10 trials will be conducted:

Trial 1- Single-Large Perturbation in Standing Trial 2- Single-Large Perturbation in Walking Trial 3- Instrumented CTSIB Trial 4- Locomotor CTSIB Trial 5- Instrumented CTSIB + Perturbations Trial 6- Locomotor CTSIB + Perturbations Trial 7- Instrumented CTSIB + Auditory Stroop Test Trial 8- Locomotor CTSIB + Auditory Stroop Test Trial 9- Instrumented CTSIB + Perturbations + Auditory Stroop Test Trial 10- Locomotor CTSIB + Perturbations + Auditory Stroop Test

Two different treadmill perturbations will be applied in addition to the Instrumented CTSIB and UHLSINT: a) slip perturbations, b) continuous perturbations. An auditory stroop task will be applied in relevant trials.

All of the trials will be performed in CAREN High-End Systems (Motek Medical BV, Amsterdam, The Netherlands) which is a motion capture system that is equipped with a treadmill mounted on a 6 degree of freedom motion base, a 360º dome-shaped virtual reality (VR) screen, and a marker-based movement analysis system.

ELIGIBILITY:
Inclusion Criteria:

* Young adults who: a) aged between 18 to 35 years old and, b) have never been diagnosed with somatosensory, visual, and vestibular deficits as reported by the participants, will be invited to participate. Community-dwelling older adults who: a) are 65 years old and over and, b) have not fallen in the last 12 months will also be invited to participate.

Exclusion Criteria:

* having had serious lower extremity injuries or operations in the past year,
* having any neurological (stroke, epilepsy, Parkinson's disease, etc.), sensory (i.e. peripheral neuropathy, diminished sense of pain, etc.) or motor disorder that can interfere with the results of the study
* Diagnosed vascular, respiratory, cardiac, orthopedic, or other disorders that affect the subject's ability to exercise safely,
* Medication affecting exercise tolerance. Additionally, based on the CAREN High-End Systems contraindications and risk factors the following exclusion criteria will be applied to the participants: a) a body weight higher than the 135 kg, b) an inability to properly adjust the harness to the respective body part due to pregnancy, colostomy bags, skin lesions that cannot be protected appropriately and any other reason that prevents a proper, pain-free adjustment of the harness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy young and older adults
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2024-10-07 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Instrumented CTSIB | Baseline
  The Clinical Test of Sensory Integration and Balance (CTSIB) is a tool used to evaluate a person's sensory integration process by manipulating different sensory inputs. It assesses how well the body uses three main sensory systems-visual, vestibular, and proprioceptive inputs-to maintain postural control. Six conditions are included in the test, each progressively altering the availability of sensory information:
  Condition 1: Eyes Open, Firm Surface Condition 2: Eyes Closed, Firm Surface Condition 3: Eyes Open, Foam Surface Condition 4: Eyes Closed, Foam Surface Condition 5: Visual Conflict, Firm Surface Condition 6: Visual Conflict, Foam Surface
UHasselt Locomotor Sensory Integration Test | Baseline
  This test was developed to evaluate sensory integration in locomotion.

OTHER OUTCOMES:
Center of Mass | Baseline
  Center of mass displacement changes between the trials will be compared to achieve the aims of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasselt University, Diepenbeek, Belgium

IPD SHARING:
Plan to Share IPD: No